CLINICAL TRIAL: NCT05932836
Title: An Pancancer Study on Organoid-on-chips Technological System Based on Biopsy Samples and Its Efficacy in Predicting the Response to MFOLFOX6 Infusion in Hepatocellular Carcinoma
Brief Title: An Organoid-on-chips Technique Based on Biopsy Samples and Its Efficacy in Predicting the Response to HAI in HCC
Status: Active, not recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: DX11330
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Drug Sensitivity; Organoid-on-chips
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Malignant solid tumor biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pancancer corhor: No interventions to be administered.
  Interventions: Other: No interventions.
- Hepatocellular carcinoma patients who undergo hepatic artery infusion with mFOLFOX6: No interventions to be administered.
  Interventions: Other: No interventions.

INTERVENTIONS:
Other: No interventions. — No interventions to be administered.

SUMMARY:
This study is aimed to establish an organoid-on-chips technological system based on biopsy samples and evaluate its efficacy in predicting the response to mFOLFOX6 infusion in patients with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a two-stage, multi-center real-world observational study. In stage 1, we aim to establish the technical system of organoid-on-chips culture system based on biopsy samples from patients with malignant solid tumors including breast cancer, lung cancer, liver cancer, bile duct cancer and pancreatic cancer, et.al. In stage 2, we aim to evaluate the predicting efficacy of the established organoid-on-chips system in HCC patients who undergo hepatic artery infusion (HAI) with mFOLFOX6 (oxaliplatin 85mg/m^2, d1, HAI for 2h; calcium folinate 200mg/m^2, d1, HAI for 1h; fluorouracil 400mg/m^2, hepatic artery injection; fluorouracil 2400mg/m^2, HAI for 46h).

ELIGIBILITY:
Inclusion Criteria for stage 1:

1. Patients who need to undergo biopsy for clinically and/or pathologically diagnosed (suspected) with malignant solid tumors including breast cancer, lung cancer, liver cancer, bile duct cancer or pancreatic cancer, et.al.
2. ECOG score ≤ 2.
3. Age between 18-75 years old.

(5) Understand and sign the informed consent form.

Exclusion Criteria for stage 1：

1. Severe heart and lung dysfunction。
2. Irreversible bleeding tendency.
3. There are obvious infectious lesions or important structures that cannot be avoided along the puncture path.

Inclusion criteria for stage 2:

1. Age 18-75 years old.
2. Hepatocellular carcinoma (HCC) confirmed by pathological histology BCLC stage C or CNLC stage IIIb; or BCLC B or CNLC IIb stage HCC progressed after previous local treatment (surgery, TACE/TAE and ablation); and treated by hepatic artery infusion with mFOLFOX6.
3. At least one lesion that can be evaluated by mRECIST criteria; lesions that have undergone local treatment (TACE/TAE, ablation, radiotherapy) should not be included (unless there is progression at baseline assessment at entry, in which case it should be classified as non-target lesions/unmeasurable lesions).
4. Liver function Child-Pugh A or B level (≤8 points).
5. ECOG PS ≤ 2 points.
6. Expected survival time > 3 months.
7. Understand and sign the informed consent form.

Exclusion criteria for stage 2:

1. Patients who have had or are currently suffering from other malignant tumors (except for cured basal or squamous cell skin cancer or cervical in situ cancer);
2. White blood cell count <2.5×10^9/L or platelet count <50×10^9/L.
3. Renal dysfunction (creatinine>2mg/L).
4. Liver dysfunction (Child-Pugh≥9 points or bilirubin>75μmol/L).
5. with grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias, and grade III-IV heart failure.
6. Poor coagulation function INR>1.5, or undergoing anticoagulant therapy or known bleeding disorders.
7. Uncontrollable systemic infection.
8. Patients who underwent chemotherapy, immunotherapy, antitumor vaccines or other antitumor drugs within 2 months.
9. Complications or social environment that may cause subjects to fail to follow the study plan or even endanger patient safety.
10. Participating in another therapeutic clinical trial at the same time.
11. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens who need to undergo biopsy for malignant tumors such as breast cancer, lung cancer, liver cancer, bile duct cancer or pancreatic cancer that have been clinically and/or pathologically diagnosed.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of organoid culture of biopsy samples | 2 years
  The number of successful cases of Organoid culture divided by the number of enrolled cases
Accuracy of Organoid drug sensitivity test in predicting the response to mFOLFOX6 infusion in HCC patients with successful Organoid culture | 3 years
  The sensitivity and specificity of drug sensitivity test in patients with successful Organoid culture to predict the response mRECIST) to mFOLFOX6 infusion in HCC

SECONDARY OUTCOMES:
Accuracy of Organoid drug sensitivity test in predicting the response to mFOLFOX6 infusion in intent-to-treat HCC population | 3 years
  The sensitivity and specificity of drug sensitivity test in patients with successful Organoid culture to predict the response mRECIST) to mFOLFOX6 infusion in intent-to-treat HCC population
The predictive effect of Organoid drug sensitivity test on the survival of patients with HCC. | 4 years
  The predictive role of Organoid drug sensitivity test results and the survival period of patients with HCC receiving mFOLFOX6 infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Liangrong Shi, MD, Study Chair — Xiangya Hospital Central South Hospital
Locations (1):
- Liangrong Shi, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet